CLINICAL TRIAL: NCT05613985
Title: A Randomised, Open-Label, Multicentre Clinical Study To Evaluate The Efficacy And Safety Of Topical Applications Of the System VULNOFAST® Plus / VULNOLIGHT® In Addition To The Usual Care Versus Usual Care Alone For The Treatment Of Infected Foot Ulcers In Diabetic Patients (PHOTOFINISH)
Brief Title: PHOTOFINISH: a Clinical Study To Evaluate The Efficacy And Safety Of the System VULNOFAST® Plus/VULNOLIGHT® In Addition To The Usual Care (UC) Vs UC Alone For The Treatment Of Infected Diabetic Foot Ulcers
Acronym: PHOTOFINISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L.Molteni & C. dei F.lli Alitti-Soc. di Esercizio S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOLT-2019-01
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Infection
Keywords: Infected diabetic foot ulcer; Diabetic foot ulcer; DFU; Infected diabetic wound; Photodynamic therapy; PDT
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Open-label, randomised, two arms study to evaluate the efficacy and safety of topical application of the system VULNOFAST® plus / VULNOLIGHT® in addition to Usual Care, versus the Usual Care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Usual Care alone (Active Comparator)
  Interventions: Other: Usual Care alone
- Arm B: system VULNOFAST® plus / VULNOLIGHT® in addition to Usual Care (Experimental)
  Interventions: Device: System VULNOFAST® plus / VULNOLIGHT® in addition to Usual Care

INTERVENTIONS:
Other: Usual Care alone — Usual Care is defined as the following procedures to apply to the foot ulcer, carried out in the order in which they are listed:
  Sharp debridement (the debridement will be performed only if non-vital tissue is present), Mild washing of the whole ulcer with physiological solution, Treatment with topical antiseptic containing Iodopovidone, Covering with iodopovidone impregnated gauze while the ulcer is clinically infected (PEDIS ≥ 2) [If, during the study, PEDIS is < 2, the ulcer will be covered with nonadherent paraffin gauze].
  Treatment 2 times a week (4 treatment weeks, 8 treatments).
  Arms: Arm A: Usual Care alone
Device: System VULNOFAST® plus / VULNOLIGHT® in addition to Usual Care — System VULNOFAST® plus / VULNOLIGHT®: VULNOFAST® plus sterile solution, in combination with a red light source VULNOLIGHT®. VULNOFAST® plus and VULNOLIGHT® will be used in accordance with their Instructions for Use (IFU) and User Manual.
  Treatments 2 times a week (4 treatment weeks, 8 treatments of Usual Care and 8 treatments of system VULNOFAST® plus / VULNOLIGHT®).
  Arms: Arm B: system VULNOFAST® plus / VULNOLIGHT® in addition to Usual Care

SUMMARY:
The aim of this randomised, open-label, multicentre clinical trial is to evaluate the superiority of the treatment which foresees the addition of the system VULNOFAST® plus / VULNOLIGHT® to the Usual Care, versus the treatment with Usual Care alone, for the healing of chronic diabetic foot ulcer. VULNOFAST® plus is a sterile solution used in combination with a red light source VULNOLIGHT®. Usual Care is defined as procedures to apply to the foot ulcer, carried out in the order in which they are listed in the protocol.

DETAILED DESCRIPTION:
This study evaluates the superiority of the treatment which foresees the addition of the system VULNOFAST® plus / VULNOLIGHT® to the Usual Care, versus the treatment with Usual Care alone, for the healing of chronic diabetic foot ulcer.

Eligible patients are randomised in a 1:1 ratio to receive Usual Care and the system VULNOFAST® plus / VULNOLIGHT®, or Usual Care alone according the following scheme:

* Arm A: Usual Care alone: 2 times a week (4 treatment weeks, 8 treatments).
* Arm B: system VULNOFAST® plus / VULNOLIGHT® in addition to Usual Care: both treatments 2 times a week (4 treatment weeks, 8 treatments of Usual Care and 8 treatments of system VULNOFAST® plus / VULNOLIGHT®).

The Treatment period will be followed by a Follow up period: the study will last up to 57 days for each patient, including the screening period. Thirteen study visits are planned starting from the screening and including Treatment and Follow up periods.

All patients enrolled in this study:

* are administered with amoxicillin and clavulanic acid treatment (as background antibiotic therapy) from Visit 1 until receipt of the antibiogram. Upon receipt of the antibiogram, the Investigator decides whether or not to continue the background therapy or to treat the patient with a different antibiotic treatment, according the clinical practice in the site.
* use an appropriate off-loading system from Visit 1 to Visit 12

The primary objective is to assess clinical improvement after 2 weeks of study treatment by evaluation of the following primary endpoint:

- proportion of patients who had total bacterial load ≤ 1000 CFU/ml at Visit 5 (Visit 5 is the first visit of 3rd week of treatment), measured by punch biopsy.

The key secondary objective is also to assess clinical improvement after 4 weeks of study treatment reflected by the key secondary endpoint:

- proportion of patients who had a reduction of the target ulcer area ≥ 40% from the baseline (Visit 1) to the first follow-up visit (Visit 9) after 4 weeks of study treatment, assessed by MolecuLight i:X medical device.

Further secondary objectives are evaluated in the study, and a pharmacoeconomic analysis is foreseen.

ELIGIBILITY:
Main Inclusion Criteria:

* Able and willing to give voluntary written informed consent. The ICF, must be signed before any study-related procedures and/or assessments are performed.
* Outpatients or inpatients (male and female) of any ethnic origin, aged 18 years or over, diagnosed with type 1 or type 2 diabetes mellitus.
* Glycaemic control confirmed by a glycated haemoglobin (HbA1c) levels ≤10% (86 mmol/mol), evaluated in the 3 months before enrolment or at Visit 1.
* Fasting plasma glucose (FPG) less than 300 mg/dl.
* A chronic diabetic foot ulcer (DFU) below the malleolus, with an area ≥ 2 and ≤ 40 cm2 and with a maximum diameter/length ≤ 10 cm measured by MolecuLight i:X medical device [note: chronic wound is defined as a wound that, after the normal clinical practice, does not start healing within 4 weeks or does not heal within 8 weeks].
* A diabetic foot wound with a depth equal or higher to grade 2 according to the category "Depth/tissue loss" of PEDIS, but not involving bone, diagnosed by clinical examination.
* Presence of infected foot ulcer of grade 2 according to the category "Infection" of PEDIS, diagnosed by clinical examination.
* Able to take oral medications.
* Patients must be willing and able to comply with the protocol and study procedures.

Main Exclusion Criteria:

* Patients unable to give written informed consent.
* Females who are pregnant or lactating.
* Females who are of child bearing potential and not taking adequate contraceptive precautions are excluded from the trial. Females of child bearing potential taking acceptable contraceptive precautions can be included.
* Participation in any other clinical trial or currently receiving any other investigational product(s) within 30 days prior to Visit 1.
* Ankle brachial systolic blood pressure index < 0.5 (Winsor Index) in the infected limb.
* Ulcer probe to bone positive.
* Any surgery planned during the study period (from ICF signature to last planned follow-up visit).
* Clinical diagnosis of peripheral vascular disease (PVD) requiring percutaneous or surgical revascularization.
* Transcutaneous oximetry (TcPo2) measurement < 30 mmHg.
* Use of any antibiotics (local or systemic) within 48h before Visit 1.
* Patient for whom punch biopsy is contraindicated.
* Patients that cannot take amoxicillin and clavulanic acid (background antibiotic therapy) at the dosage stated in the protocol and according to the current Summary of Product Characteristics (SPC).
* Patients that cannot be treated with topical antiseptic containing Iodopovidone and/or with iodopovidone impregnated gauze according to the contraindication available in the current Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the ulcer after 2 weeks of study treatment by evaluation of the following primary endpoint: | Visit 5 is the first visit of 3rd week of treatment.
  Proportion of patients who had total bacterial load ≤ 1000 CFU/ml at Visit 5, measured by punch biopsy.

SECONDARY OUTCOMES:
The key secondary objective is to evaluate the ulcer after 4 weeks of study treatment by evaluation of the following endpoint: | Visit 9 is after 4 weeks of study treatment
  Proportion of patients who had a change of the target ulcer area ≥ 40% from the baseline (Visit 1) to the first follow-up visit (Visit 9) after 4 weeks of study treatment, assessed by MolecuLight i:X medical device.

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - U.O.C. Diabetologia e Malattie Metaboliche, Ospedale San Donato, Arezzo
  - Unit Piede Diabetico, SODc Diabetologia e Malattie del Metabolismo, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Centro di Assistenza Vulnologica, Ospedale Villa Scassi, Genova
  - Unità di Diabetologia, Endocrinologia e Malattie Metaboliche, IRCSS Centro Cardiologico Monzino, Milan
  - U.O. Malattie Endocrine del Ricambio e della Nutrizione, Azienda Ospedaliero-Universitaria Policlinico Giaccone, Palermo
  - Dipartimento di Endocrinologia e Malattie Metaboliche, Centro Piede Diabetico, Ospedale S. Maria della Misericordia, Perugia
  - SOS Diabetologia, Presidio Ospedaliero San Jacopo, Pistoia